CLINICAL TRIAL: NCT05990842
Title: "Antibiotic Prophylaxis in Clean Soft Tissue Hand Surgery Among a Population in a Developing Country: A Randomized, Parallel, Triple-Blind, Placebo-Controlled Clinical Trial"
Brief Title: "Enhancing Surgical Safety in Developing Nations: Investigating Antibiotics' Role in Hand Surgeries."
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marcos Felipe Marcatto de Abreu (Other)
Responsible Party: Sponsor-Investigator, Marcos Felipe Marcatto de Abreu, Medical Doctor, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 57490822.9.0000.5404
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Soft Tissue Injuries
Keywords: antibiotic prophylaxis; hand surgery; orthopedic surgery; postoperative care; surgical wound infection; developing country
MeSH Terms: conditions — Soft Tissue Injuries; Surgical Wound Infection | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antibiotic prophylaxis (Experimental)
  Interventions: Drug: Antibiotic
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Antibiotic — the individual will receive 1 dose of antibiotic during anesthetic induction
  Arms: antibiotic prophylaxis
Other: placebo — the individual will receive 10 ml of saline during anesthetic induction
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to compare the use of antibiotics with no use in people undergoing soft tissue hand surgery in developing countries.

The main question it aims to answer is:

• Is an antibiotic necessary for this type of surgery in this population? Researchers will compare a group of patients who receives antibiotics during the surgical procedure with a group who receives no antibiotics to see if infection rates are the same.

ELIGIBILITY:
Inclusion Criteria:

* individuals with clean soft tissue conditions of the upper limb requiring surgery

Exclusion Criteria:

* abandonment of treatment
* ASA > 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-08-08 (Estimated); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-09-08 (Estimated)

PRIMARY OUTCOMES:
Surgical wound infection | 30 days
  CDC protocol for surgical wound infection surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Marcos M de Abreu, MD, Principal Investigator — University of Campinas, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all data will be made available, with the exception of the name of the participant
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 30 days after study publication
Access Criteria: peer reviewer of a scientific magazine